CLINICAL TRIAL: NCT01877278
Title: Wearable Pulsed Electromagnetic Fields Device in Knee Osteoarthritis Patients: a Double Blinded, Randomized Clinical Trial
Brief Title: Wearable Pulsed Electromagnetic Fields Device in Knee Osteoarthritis: Double Blinded, Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Gianfilippo Bagnato, Professore ordinario, University of Messina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11262
Record Dates: First submitted 2013-06-11; First posted 2013-06-13 (Estimated); Results first posted 2015-02-09 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-01

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Pulsed electromagnetic fields; Device; Pain; Pressure algometry
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- active (Active Comparator): Group wearing the active device emitting pulsed electromagnetic fileds
  Interventions: Device: Wearable pulsed electromagnetic fields
- placebo (Placebo Comparator): Group wearing the device non-emitting pulsed electromagnetic fileds
  Interventions: Device: Wearable pulsed electromagnetic fields

INTERVENTIONS:
Device: Wearable pulsed electromagnetic fields
  Other Names: actipatch

SUMMARY:
The aim of the study is to evaluate the efficacy of a wearable device using pulse electromagnetic fields on pain intensity reduction, measured by visual analogue score (VAS) and Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), in patients affected by osteoarthritis Secondary aim is the evaluate the effect on knee effusion reduction, when present and to evaluate pain intensity changes corrected by pain threshold measured by pressure algometry.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of primary OA of the knee according to the ACR criteria, including radiologic evidence of OA
* age >40 years
* symptomatic disease for at least 6 months prior to enrollment
* persistent pain despite receiving the maximum tolerated doses of conventional medical therapy, including acetaminophen (4 gm/day) and/or a nonsteroidal antiinflammatory drug (NSAID), with persistent pain defined as a minimum mean score of 25 mm on the visual analog scales (VAS) for global pain (0-100-mm range for each) daily pain during the month prior to study enrollment
* ability to attend followup appointments

Exclusion Criteria:

* secondary causes of OA
* local or systemic infection
* diabetes mellitus
* systemic arthritis
* allergy to anesthetic agent or contrast material
* coagulopathy
* anticoagulant therapy
* had previous IA steroid injection
* avascular necrosis of bone
* patients who are on specific OA pharmacological therapy (NSAIDS, opioids) for more than 2 weeks prior enrollment

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gianfilippo Bagnato, Professor, Study Chair — University of Messina; Gianfilippo Bagnato, MD, Principal Investigator — University of Messina
Locations (1):
- Reumatologia, Dipartimento di medicina clinica e sperimentale, Università degli studi di Messina, AOU G. Martino, Messina, Messina, Italy

REFERENCES:
- [Background] Trock DH, Bollet AJ, Dyer RH Jr, Fielding LP, Miner WK, Markoll R. A double-blind trial of the clinical effects of pulsed electromagnetic fields in osteoarthritis. J Rheumatol. 1993 Mar;20(3):456-60. PMID 8478852
- [Background] Thamsborg G, Florescu A, Oturai P, Fallentin E, Tritsaris K, Dissing S. Treatment of knee osteoarthritis with pulsed electromagnetic fields: a randomized, double-blind, placebo-controlled study. Osteoarthritis Cartilage. 2005 Jul;13(7):575-81. doi: 10.1016/j.joca.2005.02.012. PMID 15979009
- [Background] Pipitone N, Scott DL. Magnetic pulse treatment for knee osteoarthritis: a randomised, double-blind, placebo-controlled study. Curr Med Res Opin. 2001;17(3):190-6. doi: 10.1185/0300799039117061. PMID 11900312
- [Derived] Bagnato GL, Miceli G, Marino N, Sciortino D, Bagnato GF. Pulsed electromagnetic fields in knee osteoarthritis: a double blind, placebo-controlled, randomized clinical trial. Rheumatology (Oxford). 2016 Apr;55(4):755-62. doi: 10.1093/rheumatology/kev426. Epub 2015 Dec 24. PMID 26705327

RESULTS

PARTICIPANT FLOW:
Groups:
- Active: emitting group
  Wearable pulsed electromagnetic fields
- Placebo: non emitting device
  Wearable pulsed electromagnetic fields
Period: Overall Study
Arm/Group | Active | Placebo
Started | 33 | 33
Completed | 30 | 30
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.6 (11.9) | 66.9 (10) | 67.7 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 42
  Male | 9 | 9 | 18
Region of Enrollment [Number; unit: participants]
  Italy | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pain Perception Measured on Visual Analog Score (VAS) at Week 4
Description: visual analogue scale (VAS) is a validated self report instrument assessing self report pain intensity Possible scores ranges:from 0 (no pain) to 100 (the maximum of pain)
Time Frame: baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active | Placebo
Number analyzed (Participants) | 30 | 30
units on a scale
  VAS (baseline) | 67 (16) | 63.6 (15)
  VAS (after 1 month of treatment) | 50 (16) | 61 (15)
Statistical Analysis 1: Comparison: Active; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

2. Primary Outcome: Changes From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) at Week 4
Description: Multi-item questionnaire used to assess pain, stiffness, and physical function in patients with knee osteoarthritis.
  The WOMAC consists of 24 items divided into 3 subscales:
  Pain (5 items), Stiffness (2 items) and Physical Function (17 items). Score Range: On the Likert Scale version, the scores are summed for items in each subscale, with possible ranges as follows: pain=0-50, stiffness=0-20, physical function=0-170. A total WOMAC score is created by summing the items for all three subscales. A higher score represents a worse outcome.
Time Frame: baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active | Placebo
Number analyzed (Participants) | 30 | 30
units on a scale
  WOMAC total (baseline) | 136 (49) | 129.2 (40.8)
  WOMAC total (4 weeks) | 111 (48) | 126 (39)
Statistical Analysis 1: Comparison: Active; Test type: Superiority or Other; p = 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Active | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No